CLINICAL TRIAL: NCT06721767
Title: The Multidisciplinary and Multiparametric Monitoring of Patients With Inflammatory Bowel Diseases: the Experience of the Reference Center of the Emilia-Romagna
Brief Title: Monitoring of Patients With Inflammatory Bowel Diseases: the Experience of the Reference Center of the Emilia-Romagna
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: OMNIA
Record Dates: First submitted 2024-11-28; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: IBD - Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is observational with descriptive purposes, aimed at enhancing and deepening current knowledge and providing a foundation for future studies. Specifically, it seeks to identify predictive factors for aggressive disease progression, the development of frailty, the need for surgery and post-surgical outcomes, the development of neoplasia, the assessment of drug safety, and the quality of life in relation to medications or post-surgery.

DETAILED DESCRIPTION:
The total duration of the study is expected to be 10 years. Partial analyses will be conducted during the study for data publication. The clinical data required by the protocol will be collected in a pseudonymized form by personnel designated by the Principal Investigator in an electronic Case Report Form (CRF).

Analysis Methodology:

Descriptive statistical analyses will be used to describe the characteristics of the enrolled patient sample. Continuous variables will be summarized using means, standard deviations, minimum and maximum values, and percentiles. Discrete or nominal variables will be reported as absolute frequencies and relative percentage frequencies.

To study the predictive factors for disease progression, development of frailty, need for surgery, etc. (primary objectives), multivariate models (logistic regression analysis) will be used, and Odds Ratios with 95% confidence intervals (OR - CI 95%) will be calculated.

The calculation of frequencies and the estimation of event incidences, such as drug resistance, development of comorbidities, extraintestinal manifestations, and other observed episodes/events (secondary objectives) will be accompanied by their respective 95% confidence intervals (CI 95%). Analyses may focus on subcohorts of patients with different demographic and clinical-diagnostic characteristics to evaluate their varying risk probabilities.

Data will be processed using IBM SPSS statistical software (version 25.0).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age > 14 years
* Diagnosis of inflammatory bowel disease (Crohn's Disease, Ulcerative Colitis, Indeterminate Colitis, Microscopic Colitis) according to ECCO guidelines
* Having undergone at least one outpatient visit and/or hospitalization at the Regional Reference Center for IBD "Massimo Campieri"
* Acquisition of written informed consent from the patient and/or both parents/legal guardian

Exclusion Criteria:

- None

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of adult patients with IBD being followed at the Regional Reference Center "Massimo Campieri," which includes the General Surgery Unit and the IBD Specialties Unit of IRCCS AOUBO for the management of intestinal and extraintestinal conditions. Enrollment will take place in the IBD Specialties Unit during follow-up outpatient visits, hospital admissions, or through a phone/email invitation conducted by staff affiliated with the Unit.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2034-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with aggressive disease progression. | Baseline; through study completion, an average of 8 year
  Occurrence, at least once during the natural history of the patient's disease, of one or more characteristics of aggressiveness, namely:
  * Immunosuppressive/biotechnology/small molecule therapy due to failure of conventional therapy or severe disease
  * Surgery due to failure of medical therapy or the onset of complications such as strictures or fistulas
  * Endoscopic recurrence of disease post-surgery
  * Hospitalization for severe disease or the onset of complications
Percentage of fragility patients. | Baseline; through study completion, an average of 8 year
  Presence of one or more characteristics of frailty, namely:
  * Polypharmacy (defined as the need to take at least one other medication for a condition other than inflammatory bowel disease)
  * Short bowel syndrome post-surgery (defined as a small intestine length, measured from the duodenojejunal flexure, less than 200 cm) requiring supplemental enteral/parenteral nutrition
  * Osteoporosis (defined as bone mineral density - BMD - with a T-score less than -2.5) with or without pathological fractures
  * One or more extraintestinal manifestations (EIMs)
Percentage of patients with the development of comorbidities. | Baseline; through study completion, an average of 8 year
  Presence or absence of other comorbidities.
Percentage of patients with extraintestinal manifestations (EIMs). | Baseline; through study completion, an average of 8 year
  Presence or absence of extraintestinal manifestations.
Percentage of patients who underwent surgery. | Baseline; through study completion, an average of 8 year
  Number of surgical interventions for luminal disease (defined as disease affecting one or more segments of the gastrointestinal tract).
  Number of surgical interventions for perianal disease (defined as the presence of perianal fistulas, abscesses, ulcers, and anal strictures).
Percentage of patients with post-surgical complications. | Baseline; through study completion, an average of 8 year
  Presence of one or more of the following elements:
  * Early complication (< 30 days) or late complication (> 30 days) post-surgery
  * Development of short bowel syndrome (defined as a small intestine length, measured from the duodenojejunal flexure, less than 200 cm) post-surgery (if Crohn's disease)
  * Need for major therapy post-surgery
Percentage of patients with a diagnosis of neoplastic disease. | Baseline; through study completion, an average of 8 year
  Presence and typing of the neoplasm, confirmed by instrumental/radiological findings and histological verification.
Percentage of patients with drug resistance. | Baseline; through study completion, an average of 8 year
  Failure:
  * Primary
  * Secondary
  * Primary failure refers to the lack of efficacy after the induction phase, while secondary failure refers to the loss of efficacy after initial benefit.

SECONDARY OUTCOMES:
Percentage of patients with an adverse drug reaction. | Baseline; through study completion, an average of 8 year
  Occurrence of adverse drug reactions classified by:
  * Type of adverse drug event
  * Severity of the adverse event according to CTCAE 5.0
IBD-Q score | Baseline; through study completion, an average of 8 year
  Inflammatory Bowel Disease - Questionnaire (validated questionnaire).
Percentage of gastrointestinal and non-gastrointestinal infections. | Baseline; through study completion, an average of 8 year
  Assessment of the presence or absence of infections, including the type of infection/etiology if available, diagnosed through specific serology or culture tests.
Overall survival (OS) after the diagnosis of neoplastic/infectious disease. | Baseline; through study completion, an average of 8 year
  Days elapsed between the date of diagnosis of neoplasia/infection and the date of death.
Evaluation of the ergonomics of the tool and its data analysis performance. | Baseline; through study completion, an average of 8 year
  Introduction of a specific VAS scale for evaluating performance.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rizzello, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy